CLINICAL TRIAL: NCT04399070
Title: Effect of S-ketamine on Depressed Patients Undergoing Electroconvulsive Therapy-a Randomized, Double-blind, Controlled Clinical Study
Brief Title: The Effect of S-ketamine for Patients Undergoing Electroconvulsive Therapy (ECT)
Acronym: ECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yan Qiu (Other)
Responsible Party: Sponsor-Investigator, Yan Qiu, Attending Physician, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: West China Hospital Anes
Record Dates: First submitted 2020-05-08; First posted 2020-05-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Depression, Bipolar; Depression, Unipolar; Major Depressive Disorder; Manic-Depressive - Now Depressed
Keywords: Electroconvulsive therapy; Depression; S-ketamine
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder; Depressive Disorder, Major; Depression | interventions — Esketamine; Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propofol group (Placebo Comparator): patients were treated with propofol 1 mg/kg and saline bolus infusion before ECT
  Interventions: Drug: saline
- Ketamine group (Active Comparator): patients were treated with propofol 1 mg/kg and ketamine 0.5 mg/kg bolus infusion before ECT
  Interventions: Drug: ketamine
- S-ketamine group (Experimental): patients were treated with propofol 1 mg/kg and S-ketamine 0.25 mg/kg bolus infusion before ECT
  Interventions: Drug: S-ketamine

INTERVENTIONS:
Drug: S-ketamine — The depression patients received propofol and S-ketamine before ECT
  Arms: S-ketamine group
Drug: ketamine — The depression patients received propofol and ketamine before ECT
  Arms: Ketamine group
Drug: saline — The depression patients received propofol and saline before ECT
  Arms: Propofol group

SUMMARY:
This study will determine the effectiveness and safety of S-Ketamine in depression patients undergoing electroconvulsive therapy.

DETAILED DESCRIPTION:
Nowadays, depression has become one of the serious mental diseases that affect human's life. With the acceleration of life pace and social pressure, the incidence of depression is increasing year-on-year. According to the statistics of the WHO, by 2017, there were more than 300 million people suffering from depression, accounting for 4.4% of the global population. Depression is highly related to suicide, which is an important reason for suicidal intention and attempt. It has been demonstrated that the incidence of suicide associated with major depression was as high as 15%. The main characteristic of depression is significant and lasting depression, which is caused by the decrease of monoamine transmitters (including dopamine, 5-HT, et al.) related to mood. In the past, antidepressants mainly relied on increasing or reducing the metabolism of transmitters, but these drugs usually took weeks or even months to take effect, and although the symptoms of depression were relieved within weeks after the start of treatment, they were still not ideal in the long term. Therefore, the drug treatment of depression is not optimistic.

Electroconvulsive therapy (ECT), as the first biological therapy introduced into psychiatry, has been improving with the progress of technology and equipment. More studies show that ECT is a safe and effective treatment, and the treatment of severe depression is the first choice in some cases. However, cognitive dysfunction, relapse tendency and related safety after ECT need further study.

Short acting sedatives and muscle relaxants before ECT can minimize the fear and muscle pain caused by ECT induced seizures. Previous sedatives used include propofol, mesaclopidol, thiopental and ketamine. Ketamine can be used for ECT anesthesia in patients with depression because of its good epileptic characteristics and prevention of cognitive dysfunction after ECT. More evidences reveal ketamine has strong antidepressant effect and reduces suicide of patients with treatment-resistant depression or mania. The low dose of ketamine can take effect within one hour, produce rapid antidepressant effect, and can play a role in more than 70% of patients with refractory depression. In addition, even a single intravenous injection of ketamine can effectively reduce the symptoms of depression within 24-72 hours, and may have synergistic antidepressant effect when combined with ECT. Although ketamine is considered to have a significant antidepressant effect in patients with depression, its application in mental disorders remains to be further explored because it may aggravate mental symptoms. However, some studies also found that ketamine did not significantly improve the effect of ECT on depression compared with other anesthetics.

Esketamine is the isomer of ketamine, which mainly acts on NMDA receptor of glutamate and its affinity to the receptor is 3-4 times that of ketamine, therefore it has stronger effect. Evidence suggests that esketamine can regulate NMDA receptor, increase the release of various neurotransmitters, improve the depression of patients, and repair the damaged neurons to improve the neuronal connections in the brain. As an anesthetic, the potency of esketamine is two times higher than ketamine, three times higher than R-ketamine, and its drug metabolism time is shorter, and the related side effects are also significantly reduced. Conseuqently, it has been widely used as an anesthetic in some countries. The efficacy and safety of esketamine nasal spray as a rapid and effective antidepressant in the treatment of patients with refractory depression have been confirmed. However the effect of intravenous esketamine as an anesthetic in ECT anesthesia on patients who are depressed remains unknown. The aim of this study is to evaluate the short-term effect and safety of esketamine as a adjunctive anesthetic in routine ECT anesthesia for patients with depression.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status I-II
* diagnose depressive disorders with DSM-IV
* Without cognitive impairment
* Without ECT in past 6 months

Exclusion Criteria:

* had other comorbid psychiatric diagnoses, including schizophrenia, mania
* organic heart diseases, severe hypertension and arrhythmia
* severe hepatic and renal diseases
* severe cerebrovascular disorder or malformation, intracranial mass lesions and seizure
* glaucoma or high intraocular pressure and intra-ocular pathology
* severe haematological disease, fracture and obesity, pregnancy
* severe respiratory tract disease or difficult ventilation or incubation
* had pre-existing neurological disease or cognitive impairment
* allergy to anesthetics
* drugs abuse or alcohol addiction
* family history of malignant hyperthemia
* refuse to participate in this trial, had taken part in other clinical trial and with less education and couldn't understand the content of questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale-17 scores | the 1 day after the last ECT
  the patients' depression were evaluated with Hamilton Depression Scale with 17 questions after ECT. The scores ranged 0-68, and <7 were normal, the higher the score means more serious disease.
Montgomery-Asberg Depression Rating Scale scores | the 1 day after the last ECT
  the patients' depression were evaluated with Montgomery-Asberg Depression Rating Scale scores after ECT. The scores ranged 0-60, and <17 were normal, the higher the score means more serious disease.

SECONDARY OUTCOMES:
Hamilton Depression Scale-17 scores | baseline (before first ECT)
  the patients' depression were evaluated with Hamilton Depression Scale with 17 questions before ECT. The scores ranged 0-68, and <7 were normal, the higher the score means more serious disease.
Hamilton Depression Scale-17 scores | one week after the first ECT
  the patients' depression were evaluated with Hamilton Depression Scale with 17 questions after ECT. The scores ranged 0-68, and <7 were normal, the higher the score means more serious disease.
Hamilton Depression Scale-17 scores | one month after the last ECT
  the patients' depression were evaluated with Hamilton Depression Scale with 17 questions after ECT. The scores ranged 0-68, and <7 were normal, the higher the score means more serious disease.
Montgomery-Asberg Depression Rating Scale scores | baseline (before first ECT)
  the patients' depression were evaluated with Montgomery-Asberg Depression Rating Scale scores before ECT. The scores ranged 0-60, and <17 were normal, the higher the score means more serious disease.
Montgomery-Asberg Depression Rating Scale scores | one week after the first ECT
  the patients' depression were evaluated with Montgomery-Asberg Depression Rating Scale scores after ECT. The scores ranged 0-60, and <17 were normal, the higher the score means more serious disease.
Montgomery-Asberg Depression Rating Scale scores | one month after the last ECT
  the patients' depression were evaluated with Montgomery-Asberg Depression Rating Scale scores after ECT. The scores ranged 0-60, and <17 were normal, the higher the score means more serious disease.
Mini-mental State Examination scores | baseline (before first ECT)
  the patients' cognitive function were evaluated with Mini-mental State Examination scores before ECT. The scores ranged 0-30, and 27-30 were normal, the lower the score means more serious disease.
Mini-mental State Examination scores | one week after the first ECT
  the patients' cognitive function were evaluated with Mini-mental State Examination scores after ECT. The scores ranged 0-30, and 27-30 were normal, the lower the score means more serious disease.
Mini-mental State Examination scores | the 1 day after the last ECT
  the patients' cognitive function were evaluated with Mini-mental State Examination scores after ECT. The scores ranged 0-30, and 27-30 were normal, the lower the score means more serious disease.
Mini-mental State Examination scores | one month after the last ECT
  the patients' cognitive function were evaluated with Mini-mental State Examination scores after ECT. The scores ranged 0-30, and 27-30 were normal, the lower the score means more serious disease.
suicide | times of symptomatic episodes from first ECT up to one month after last ECT
  adverse events
Mean heart rate before ECT | 5 minutes before each ECT
  patients' vital sign
Mean heart rate after ECT | 5 minutes after patients emergency from each ECT
  patients' vital sign
Mean Arterial Pressure before ECT | 5 minutes before each ECT
  patients' vital sign
Mean Arterial Pressure after ECT | 5 minutes after patients emergency from each ECT
  patients' vital sign
Mean time for return of spontaneous respiration after ECT | from end of ECT to return of spontaneous respiration after each ECT
  time for return of spontaneous respiration after ECT
Mean emergency time after ECT | from end of ECT to eye opening or following commands after each ECT
  patients' recovery time after ECT
Mean seizure duration during ECT | from end of electrical stimulus to clonic movements in the right lower limb during each ECT
  patients' seizure duration during ECT

OTHER OUTCOMES:
Headache | from emergency, assessed up to 24 hours after each ECT
  adverse events
Nausea and vomiting | from emergency, assessed up to 24 hours after each ECT
  adverse events
Myalgia | from emergency, assessed up to 24 hours after each ECT
  adverse events
Agitation | from emergency, assessed up to 1 hour after each ECT
  adverse events
Hallucinations | from emergency, assessed up to 3 hours after each ECT
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Guizhi Du, Doctor, Principal Investigator — West China Hospital of Sichuan University, Department of Anesthesiology
Locations (1):
- West China Hospital of Sichuan University, Department of Anesthesiology, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. Depression and other common mental disorders: Global health estimates. Geneva: World Health Organization. 2017.
- [Background] Ribeiro JD, Huang X, Fox KR, Franklin JC. Depression and hopelessness as risk factors for suicide ideation, attempts and death: meta-analysis of longitudinal studies. Br J Psychiatry. 2018 May;212(5):279-286. doi: 10.1192/bjp.2018.27. Epub 2018 Mar 28. PMID 29587888
- [Background] Rong C, Park C, Rosenblat JD, Subramaniapillai M, Zuckerman H, Fus D, Lee YL, Pan Z, Brietzke E, Mansur RB, Cha DS, Lui LMW, McIntyre RS. Predictors of Response to Ketamine in Treatment Resistant Major Depressive Disorder and Bipolar Disorder. Int J Environ Res Public Health. 2018 Apr 17;15(4):771. doi: 10.3390/ijerph15040771. PMID 29673146
- [Background] Kellner CH, Husain MM, Knapp RG, McCall WV, Petrides G, Rudorfer MV, Young RC, Sampson S, McClintock SM, Mueller M, Prudic J, Greenberg RM, Weiner RD, Bailine SH, Rosenquist PB, Raza A, Kaliora S, Latoussakis V, Tobias KG, Briggs MC, Liebman LS, Geduldig ET, Teklehaimanot AA, Lisanby SH; CORE/PRIDE Work Group. Right Unilateral Ultrabrief Pulse ECT in Geriatric Depression: Phase 1 of the PRIDE Study. Am J Psychiatry. 2016 Nov 1;173(11):1101-1109. doi: 10.1176/appi.ajp.2016.15081101. Epub 2016 Jul 15. PMID 27418379
- [Background] Kellner CH, Husain MM, Knapp RG, McCall WV, Petrides G, Rudorfer MV, Young RC, Sampson S, McClintock SM, Mueller M, Prudic J, Greenberg RM, Weiner RD, Bailine SH, Rosenquist PB, Raza A, Kaliora S, Latoussakis V, Tobias KG, Briggs MC, Liebman LS, Geduldig ET, Teklehaimanot AA, Dooley M, Lisanby SH; CORE/PRIDE Work Group. A Novel Strategy for Continuation ECT in Geriatric Depression: Phase 2 of the PRIDE Study. Am J Psychiatry. 2016 Nov 1;173(11):1110-1118. doi: 10.1176/appi.ajp.2016.16010118. Epub 2016 Jul 15. PMID 27418381
- [Background] Fond G, Bennabi D, Haffen E, Brunel L, Micoulaud-Franchi JA, Loundou A, Lancon C, Llorca PM, Auquier P, Boyer L. A Bayesian framework systematic review and meta-analysis of anesthetic agents effectiveness/tolerability profile in electroconvulsive therapy for major depression. Sci Rep. 2016 Jan 25;6:19847. doi: 10.1038/srep19847. PMID 26806849
- [Background] Hashimoto K. Rapid-acting antidepressant ketamine, its metabolites and other candidates: A historical overview and future perspective. Psychiatry Clin Neurosci. 2019 Oct;73(10):613-627. doi: 10.1111/pcn.12902. Epub 2019 Jul 11. PMID 31215725
- [Background] Li DJ, Wang FC, Chu CS, Chen TY, Tang CH, Yang WC, Chow PC, Wu CK, Tseng PT, Lin PY. Significant treatment effect of add-on ketamine anesthesia in electroconvulsive therapy in depressive patients: A meta-analysis. Eur Neuropsychopharmacol. 2017 Jan;27(1):29-41. doi: 10.1016/j.euroneuro.2016.11.008. Epub 2016 Nov 28. PMID 27908572
- [Background] Erdil F, Ozgul U, Colak C, Cumurcu B, Durmus M. Effect of the Addition of Ketamine to Sevoflurane Anesthesia on Seizure Duration in Electroconvulsive Therapy. J ECT. 2015 Sep;31(3):182-5. doi: 10.1097/YCT.0000000000000225. PMID 25719444
- [Background] Kishimoto T, Chawla JM, Hagi K, Zarate CA, Kane JM, Bauer M, Correll CU. Single-dose infusion ketamine and non-ketamine N-methyl-d-aspartate receptor antagonists for unipolar and bipolar depression: a meta-analysis of efficacy, safety and time trajectories. Psychol Med. 2016 May;46(7):1459-72. doi: 10.1017/S0033291716000064. Epub 2016 Feb 12. PMID 26867988
- [Background] Wilkinson ST, Ballard ED, Bloch MH, Mathew SJ, Murrough JW, Feder A, Sos P, Wang G, Zarate CA Jr, Sanacora G. The Effect of a Single Dose of Intravenous Ketamine on Suicidal Ideation: A Systematic Review and Individual Participant Data Meta-Analysis. Am J Psychiatry. 2018 Feb 1;175(2):150-158. doi: 10.1176/appi.ajp.2017.17040472. Epub 2017 Oct 3. PMID 28969441
- [Background] Zhang K, Hashimoto K. An update on ketamine and its two enantiomers as rapid-acting antidepressants. Expert Rev Neurother. 2019 Jan;19(1):83-92. doi: 10.1080/14737175.2019.1554434. Epub 2018 Dec 4. PMID 30513009
- [Background] Sackeim HA. Modern Electroconvulsive Therapy: Vastly Improved yet Greatly Underused. JAMA Psychiatry. 2017 Aug 1;74(8):779-780. doi: 10.1001/jamapsychiatry.2017.1670. No abstract available. PMID 28658461
- [Background] Carspecken CW, Borisovskaya A, Lan ST, Heller K, Buchholz J, Ruskin D, Rozet I. Ketamine Anesthesia Does Not Improve Depression Scores in Electroconvulsive Therapy: A Randomized Clinical Trial. J Neurosurg Anesthesiol. 2018 Oct;30(4):305-313. doi: 10.1097/ANA.0000000000000511. PMID 29847468
- [Background] Zheng W, Li XH, Zhu XM, Cai DB, Yang XH, Ungvari GS, Ng CH, Ning YP, Hu YD, He SH, Wang G, Xiang YT. Adjunctive ketamine and electroconvulsive therapy for major depressive disorder: A meta-analysis of randomized controlled trials. J Affect Disord. 2019 May 1;250:123-131. doi: 10.1016/j.jad.2019.02.044. Epub 2019 Feb 18. PMID 30852364
- [Background] Daly EJ, Singh JB, Fedgchin M, Cooper K, Lim P, Shelton RC, Thase ME, Winokur A, Van Nueten L, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine Adjunctive to Oral Antidepressant Therapy in Treatment-Resistant Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Feb 1;75(2):139-148. doi: 10.1001/jamapsychiatry.2017.3739. PMID 29282469
- [Background] Popova V, Daly EJ, Trivedi M, Cooper K, Lane R, Lim P, Mazzucco C, Hough D, Thase ME, Shelton RC, Molero P, Vieta E, Bajbouj M, Manji H, Drevets WC, Singh JB. Efficacy and Safety of Flexibly Dosed Esketamine Nasal Spray Combined With a Newly Initiated Oral Antidepressant in Treatment-Resistant Depression: A Randomized Double-Blind Active-Controlled Study. Am J Psychiatry. 2019 Jun 1;176(6):428-438. doi: 10.1176/appi.ajp.2019.19020172. Epub 2019 May 21. PMID 31109201
- [Background] Canuso CM, Singh JB, Fedgchin M, Alphs L, Lane R, Lim P, Pinter C, Hough D, Sanacora G, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of Symptoms of Depression and Suicidality in Patients at Imminent Risk for Suicide: Results of a Double-Blind, Randomized, Placebo-Controlled Study. Am J Psychiatry. 2018 Jul 1;175(7):620-630. doi: 10.1176/appi.ajp.2018.17060720. Epub 2018 Apr 16. PMID 29656663